CLINICAL TRIAL: NCT04208386
Title: A Phase 1, Single-Dose, Open-Label, Parallel-Group Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of JNJ-73763989
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on JNJ-73763989
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108708; 73763989HPB1002 (Other: Janssen Sciences Ireland UC); 2019-003083-51 (EudraCT Number)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: Group 1 (Experimental): Participants with liver cirrhosis with moderate hepatic impairment will receive single subcutaneous (SC) injection of JNJ-73763989 on Day 1 under fasted condition.
  Interventions: Drug: JNJ-73763989
- Part A: Group 2 (Experimental): Participants with normal liver function with no liver cirrhosis will receive single SC injection of JNJ-73763989 on Day 1 under fasted condition.
  Interventions: Drug: JNJ-73763989
- Part B: Group 3 (optional) (Experimental): Participants with liver cirrhosis with mild hepatic impairment will receive single SC injection of JNJ-73763989 on Day 1 under fasted condition.
  Interventions: Drug: JNJ-73763989
- Part B: Group 4 (optional) (Experimental): Participants with liver cirrhosis with severe hepatic impairment will receive SC injection of JNJ-73763989 on Day 1 under fasted condition.
  Interventions: Drug: JNJ-73763989

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 will be administered SC under fasted condition.

SUMMARY:
The purpose of the study is to evaluate the single-dose pharmacokinetic (PK) of JNJ-73763976 and JNJ-73763924 following a subcutaneous (SC) injection of JNJ-73763989 (JNJ-3989) in participants with liver cirrhosis and various degrees of impaired hepatic function when compared with healthy participants with normal hepatic function and no liver cirrhosis.

ELIGIBILITY:
Inclusion criteria:

* For all participants: Body mass index (BMI) between 18.0 and 38 kilogram per meter square (kg/m^2), (extremes included), and a body weight not less than 50 kilograms (kg) at screening; Woman of childbearing potential must not be pregnant; Highly effective contraceptive measures in place for female participants of childbearing potential or male participants with female partners of childbearing potential; Non-smoker or light smoker as defined per protocol
* For Healthy Participants with Normal Hepatic Function and No Liver Cirrhosis: Demographically comparable to the study groups with hepatic impairment with respect to sex, age (+/-10 years), and body weight (+/-10 kg); Participants must be in good health clinically and biologically as defined per protocol
* For Participants with Liver Cirrhosis and Moderate or Mild or Severe Hepatic Impairment: Must have a total Child-Pugh score of 5 or 6, inclusive (mild); or 7 to 9, inclusive (moderate); or 10 to 15, inclusive (severe) as determined by the investigator; Must have liver cirrhosis with fibro scan readout greater than (>) 12.5 Kilopascal (kPa) as cut-off at screening
* Participants with controlled hypertension, with problems directly associated with the primary diagnosis of hepatic impairment may be included. Participants may have concurrent stable medical conditions and may be included in the study if the investigator and the sponsor consider that the condition(s) will not introduce an additional risk factor and will not interfere with the study objectives and the procedures (that is, participants with mild degenerative joint disease, controlled diabetes, controlled thyroid conditions, other conditions addressed on a case by case basis)
* Concomitant medications to treat underlying disease states or medical conditions related to hepatic impairment are allowed

Exclusion Criteria:

* History of/or current clinically significant medical illness that could interfere with the interpretation of the study results.
* Known allergies, hypersensitivity, or intolerance to JNJ-3989 or its excipients.
* History of drug or alcohol abuse within 1 year before screening or positive test results at screening and Day -1.
* Blood or blood products donated or substantial loss of blood (more than 500 milliliters [mL]) within 3 months before the study starts
* Experimental drug received (including investigational vaccines) or experimental medical device used within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study intervention is scheduled.
* Evidence of infection with Human Immunodeficiency Virus (HIV)-1 and HIV-2, hepatitis A, B or C (except if sustained virologic response to HCV treatment)
* Inability to fast for 10 hours
* Signs of hepatocellular carcinoma or history of biliary obstruction within the past 2 years
* Lack of good or reasonable venous access
* Use of any disallowed therapies as per protocol
* Participants with advanced renal disease with staggered estimated glomerular filtration rate (eGFR) cutoff for increasing degree of hepatic impairment
* History of Liver transplant, gastroesophageal variceal bleeding within 6 months prior to screening, known gastric varices, uncontrolled ascites, spontaneous bacterial peritonitis within 3 months before screening
* Acute or exacerbating hepatitis, fluctuating or rapidly deteriorating hepatic function or use of any therapy known to exacerbate hepatic dysfunction within 2 weeks of study intervention administration
* Clinically significant laboratory findings except as related to hepatic impairment as defined per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of JNJ-73763989 | Up to Day 4
  Plasma concentration of oral dose of JNJ-73763989 will be reported.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 42 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Kakuda TN, Halabi A, Klein G, Sanga M, Guinard-Azadian C, Kowalik M, Nedoschinsky K, Nangosyah J, Ediage EN, Hillewaert V, Verboven P, Goris I, Snoeys J, Palmer M, Biermer M. Pharmacokinetics of JNJ-73763989 and JNJ-56136379 (Bersacapavir) in Participants With Moderate Hepatic Impairment. J Clin Pharmacol. 2023 Jun;63(6):732-741. doi: 10.1002/jcph.2214. Epub 2023 Mar 20. PMID 36786053